CLINICAL TRIAL: NCT03571737
Title: Efficacy of Lidocaine Patch in Acute Musculoskeletal Pain in the Emergency Department: A Prospective Randomized Controlled Study
Brief Title: Efficacy of Lidocaine Patch in Acute Musculoskeletal Pain in the Emergency Department
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Stahl, Jennifer, MD, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCIRB 17-001594
Record Dates: First submitted 2018-06-02; First posted 2018-06-28 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Acute Musculoskeletal Disease; Sprains; Sprains and Strains; Injuries; Emergencies; Trauma; Acute Pain
Keywords: acute pain; muscle strain; muscle sprain; injury; emergency department
MeSH Terms: conditions — Sprains and Strains; Wounds and Injuries; Emergencies; Acute Pain | interventions — Ibuprofen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibuprofen (Active Comparator): Ibuprofen 800mg every 8 hours for 3 days
  Interventions: Drug: Ibuprofen
- Ibuprofen & Lidocaine Patch 4% (Experimental): Ibuprofen 800mg every 8 hours for 3 days and Lidocaine patch 4% 1 patch applied for 12 hours then removed for 12 hours, for 3 days
  Interventions: Drug: Ibuprofen; Drug: Lidocaine Patch 4%

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen tablet
  Other Names: Motrin; Advil
Drug: Lidocaine Patch 4% — Lidocaine patch
  Other Names: Lidocaine Pain Relief Patch
  Arms: Ibuprofen & Lidocaine Patch 4%

SUMMARY:
This study evaluates the addition of a lidocaine patch to ibuprofen in the treatment of acute musculoskeletal pains. Half of the participants will get only ibuprofen for their pain, while other half will receive lidocaine patch plus the ibuprofen. After addition of the pain medications, the participants will be followed for their pain scores and return visits.

DETAILED DESCRIPTION:
Ibuprofen and other nonsteroidal antiinflammatory pain medications have been traditionally used for relief of mild to moderate acute musculoskeletal pains. However, if this medication did not work, a different modality for pain control would be added to the original regimen. In recent times, lidocaine patch has been introduced as a separate modality for pain control. This medication is thought to help by selectively inhibiting voltage-gated sodium channels in nociceptors involved in pain response. Given the separate modality, it would be prudent to see whether the addition of lidocaine patch to the ibuprofen would help relieve the pain more so than the antiinflammatory-only regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age is greater than or equal to 18 years old
* Subject is able to speak English
* Subject has chief complaint of musculoskeletal pain lasting less than or equal to 7 days
* Subject's area of greatest pain isolated to one body part
* Subject does not have prior Emergency Department visits recorded on electronic medical records for the chief complaint

Exclusion Criteria:

* Subject's age is less than 18 years old
* Subject is pregnant or breastfeeding patients
* Subject cannot speak English
* Subject has multiple traumatic injuries or injury requiring consultation with the trauma service per study facility's guidelines
* Subject has cellulitis or infection overlying the injuries
* Subject has open wound overlying the injuries
* Subject's chief complaint is caused by penetrating injury
* Subject has absolute contraindications to study medications, including anaphylaxis to lidocaine or nonsteroidal antiinflammatory drugs, history of active GI bleeding or recent coronary artery bypass graft surgery precluding nonsteroidal antiinflammatory medications, severe hepatic disease (hepatitis, cirrhosis in current chart or prior history or elevation in liver function tests to clinically significant levels in past 6 months), severe kidney disease (Creatinine clearance less than 30 milliliters or history of chronic kidney disease stage 3 or worse), congestive heart failure.
* Subject has medication contraindications such as concurrent use of medications listed: Alcuronium, Amphotericin B, Amprenavir, Atracurium, Cimetidine, Edrophonium, Enflurane, Fosphenytoin, Halothane, Nadolol, Oxprenolol, Pentazocine, Propafenone
* Subject is on class I antiarrhythmics therapy (including lidocaine, procainamide, disopyramide etc)
* Subject has injuries requiring splint/casting where patient may not be able to reach the area of greatest pain to apply and reapply the patch
* Subject has prior history of chronic pain in the affected area (defined as greater than or equal to 6 weeks of pain)
* Subject has received opioid medication in triage area or within 4 hours of initial treatment
* Subject is unable to give pain scores due to mental status
* Subject's initial numerical pain scale score of 0 (which would constitute "no pain" on the scale)
* Subject requires opiate medication or muscle relaxants (Flexeril, Valium, Tizanidine, Robaxin etc) during the initial visit to Emergency department at the discretion of the provider.
* Subjects who received less than 800 milligram oral dosage of ibuprofen in triage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-06-23 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stahl, MD, Study Director — East Carolina University
Locations (1):
- Vidant Medical Center, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibuprofen- Control: Ibuprofen 800mg every 8 hours for 3 days
  Ibuprofen: Ibuprofen tablet
- Ibuprofen & Lidocaine Patch 4%- Experimental: Ibuprofen 800mg every 8 hours for 3 days and Lidocaine patch 4% 1 patch applied for 12 hours then removed for 12 hours, for 3 days
  Ibuprofen: Ibuprofen tablet
  Lidocaine Patch 4%: Lidocaine patch
Period: Overall Study
Arm/Group | Ibuprofen- Control | Ibuprofen & Lidocaine Patch 4%- Experimental
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Ibuprofen & Lidocaine Patch 4% | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (17.3) | 36.8 (13.2) | 35.8 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 5 | 5 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23
Initial Pain Score [Mean (Standard Deviation); unit: units on a scale] — Pain score is assessed with a 10 point Likert pain scale. Scale range 0 to 10. Lower score is better outcome, higher score is worse outcome.
  Total is the combined score for both intervention groups. In this case the mean average of scores for all participants (including both intervention groups) with range score 0 to 10. Lower score is better outcome, higher score is worse outcome
  units on a scale | 6.8 (2.0) | 6.8 (2.5) | 6.8 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Numerical Pain Rating Scale
Description: Change in self-reported pain intensity level. Baseline will be prior to intervention, and change will be assessed 60 minutes after intervention. Each item is scored 0-10 (0=No pain, 10= Worst pain possible). Higher number is worse outcome while lower number is better outcome.
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ibuprofen- Control | Ibuprofen & Lidocaine Patch 4%- Experimental
Number analyzed (Participants) | 13 | 10
score on a scale | 2.9 [0.85 to 5.0] | 2.1 [.30 to 3.3]

2. Secondary Outcome: Number of Participants With a Return Visit for Same Chief Complaint
Description: Questionnaire (Yes or No) of whether a return visit to either the emergency department or primary care offices occurred within 1 week for same chief complaint from the initial visit
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen- Control | Ibuprofen & Lidocaine Patch 4%- Experimental
Number analyzed (Participants) | 13 | 10
Participants | 11 | 10

ADVERSE EVENTS:
Time Frame: From study enrollment to 7 days post-enrollment
Arm/Group | Ibuprofen- Control | Ibuprofen & Lidocaine Patch 4%- Experimental
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT03571737/Prot_001.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT03571737/SAP_002.pdf